CLINICAL TRIAL: NCT04435145
Title: The Impact of Warning Labels on Reducing College Students' Sugar-Sweetened Beverage Intake
Brief Title: Warning Labels and College Students' Sugar-Sweetened Beverage Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Cindy Leung, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HUM00153805
Record Dates: First submitted 2020-06-15; First posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Diet, Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Sugar-sweetened beverage warning label
  Interventions: Behavioral: Sugar-sweetened beverage warning label
- Control (No Intervention): No label

INTERVENTIONS:
Behavioral: Sugar-sweetened beverage warning label — A sugar-sweetened beverage warning label appropriate for the college-aged population was developed and applied to beverage stations at one large campus dining hall
  Arms: Intervention

SUMMARY:
Sugar-sweetened beverages (SSBs) are one of the few dietary items causally linked to the development of obesity and chronic disease. SSB consumption among young adults are particularly concerning, because of the high levels of consumption and the influence of disease risk in later life. College students, particularly freshmen, are a captive audience when it comes to dietary consumption because many of them consume their meals in residential dining halls. We are currently working with Michigan Dining to implement warning labels on SSB fountain dispensers to examine whether carefully tailored signage could alter beverage choices of college students. The current study aims to assess changes in dietary intake before and after the labels are posted, in a representative sample of University of Michigan students who eat at residential dining halls.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled student at the University
* Visited one of three large dining halls at least 100 times in the first 1.5 months of the academic year

Exclusion Criteria:

-

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1067 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Beverage Intake Questionnaire-15 | Four months
  The primary outcome is the mean servings of sugar-sweetened and non-sugar-sweetened beverages consumed in the past 30 days, as measured by a validated questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leung CW, Wolfson JA, Hsu R, Soster K, Mangan S, Falbe J. Warning Labels Reduce Sugar-Sweetened Beverage Intake among College Students. J Nutr. 2021 Jan 4;151(1):179-185. doi: 10.1093/jn/nxaa305. PMID 33245125